CLINICAL TRIAL: NCT04237376
Title: Chronic HBV Infection in Pregnant Women Taking TAF to Prevent Mother-to-child Transmission in the Third Trimester: a Multicenter, Prospective Study
Brief Title: Chronic HBV Infection in Pregnant Women Taking TAF to Prevent Vertical Transmission
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New Discovery LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017ZX10201201-001
Record Dates: First submitted 2019-12-21; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis B, Chronic; Pregnancy Related
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; Tenofovir; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Treatment Arm A: CHB Mothers treated with TAF during Pregnancy: 120 pregnant women with double positive HBsAg and HBeAg and HBV DNA levels ≥ 2 × 10^6 IU/mL were recruited from all four treatment centers. Mothers were enrolled and observed from gestational week 24-28 until postpartum week 28, and treated with TAF (25mg oral daily) from gestational week 28 until delivery (if the liver function is significantly abnormal after delivery, that is, ALT ≥ 5 × Upper Limit of Normal (ULN), the oral antiviral drug can be continued according to the wishes of the pregnant woman and the test results). All babies were given 3 HBV vaccines (0, 1, 6) and 1 routine Hepatitis B immunoglobin (HBIG) after birth. All babies were followed up to 2 years. According to the mother's wishes, if the mother agrees to collect breast milk and determine TAF concentration, breast milk was collected every day, and continuously collected 5-7 days for TAF concentration measurement. The time of last TAF dose taken as well as the time between milk collection and delivery was recorded.
  Interventions: Drug: Tenofovir Alafenamide 25 MG
- Comparative Arm C: CHB Pregnant Mothers: This arm C consists of 360 cases of pregnant women with HBsAg and HBeAg double-positive, and HBV DNA level ≥ 2 × 10^6 IU/mL. The mothers in this historical cohort did not receive any antiviral treatment during their pregnancy. All cases of pregnant mothers in this arm were extracted from the four treatment centers involved in this study: Beijing You'an Hospital, Capital Medical University, Fourth Hospital Affiliated to Harbin Medical University, Third Hospital of Qinhuangdao, and Tongliao Infectious Disease Hospital. All babies received 3 doses of HBV vaccine (0, 1, 6) and 1 dose of HBIG after birth.
- Comparative Arm B: CHB Pregnant Mothers treated with TDF: This retrospective cohort arm B consists of 120 cases of pregnant women with double-positive HBsAg and HBeAg and HBV DNA levels ≥ 2 × 10^6 IU/mL. All cases of pregnant mothers in this arm were extracted from the four treatment centers involved in this study: Beijing You'an Hospital, Capital Medical University, Fourth Hospital Affiliated to Harbin Medical University, Third Hospital of Qinhuangdao, and Tongliao Infectious Disease Hospital. Pregnant mothers were treated with TDF (300mg oral daily) starting from gestational week 28 and discontinued the drug at delivery. All babies received 3 doses of HBV vaccine (0, 1, 6) and 1 dose of HBIG after birth.
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG Oral Tablet

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG — Tenofovir Alafenamide 25 mg, per oral daily was taken by CHB pregnant mothers with viral load ≥ 2 × 10^6 IU / mL from gestational week 28 to delivery of infant to prevent MTCT.
  Other Names: Vemlidy
  Groups: Treatment Arm A: CHB Mothers treated with TAF during Pregnancy
Drug: Tenofovir Disoproxil Fumarate 300 MG Oral Tablet — Tenofovir Disoproxil Fumarate 300 mg, per oral daily was taken by CHB pregnant mothers with viral load ≥ 2 × 10^6 IU / mL from gestational week 28 to delivery of infant to prevent MTCT.
  Other Names: Viread
  Groups: Comparative Arm B: CHB Pregnant Mothers treated with TDF

SUMMARY:
Mother-to-child transmission is the main route of transmission of Hepatitis B Virus (HBV) in China, and about 30% - 50% of chronic HBV carriers are infected by this. Although the current hepatitis B vaccine combined with hepatitis B immunoglobulin scheme has achieved excellent results, about 5% - 10% of infants born to chronic hepatitis B (CHB) mothers are still infected. A pregnant women's blood hepatitis B virus load ≥ 2 × 10^5 IU/mL before delivery is the main risk factor for transmission prevention failure. Two recent random controlled trial (RCT) studies have shown that the use of Tenofovir Disoproxil Fumarate (TDF) in highly viremic HBsAg positive mothers may safely reduce the rate of MTCT in comparisons between groups of TDF treated and untreated patients. Tenofovir Alafenamide (TAF) is the successor to TDF, and both drugs have a similar mechanism of action to reduce HBV DNA levels and normalize serum alanine aminotransferase (ALT) in chronic hepatitis B patients (CHB). TAF however, has a better safety profile with less adverse effects to hip and spine bone mineral density and renal function. Currently, TAF has been approved by the State Food and Drug Administration and marketed in China in December 2018. On the drug label, it has been suggested that TAF may be considered during pregnancy if necessary. However, it has not been reported whether the application of TAF in pregnant women can achieve better effects and safety in prevention of mother-to-child transmission. This prospective, triple arm, multicenter study seeks to evaluate the efficacy and safety of TAF in the prevention of mother-to-child transmission as compared to a retrospective cohort of mothers who were treated with TDF.

DETAILED DESCRIPTION:
Mother-to-child transmission is the main route of transmission of HBV in China, and about 30% - 50% of chronic HBV carriers are infected by this route. Although the current hepatitis B vaccine combined with hepatitis B immunoglobulin scheme has achieved excellent results, about 5% - 10% of transmission prevention failure still occur. More than 90% of newborns will develop chronic infection after HBV infection, and about one quarter will eventually develop cirrhosis and / or hepatocellular carcinoma, which is extremely serious. Therefore, improving and optimizing the current transmission prevention technology and program to further increase the success rate of HBV mother-to-child prevention is to reduce the transmission and prevalence of HBV in China, reduce the burden of hepatitis B disease, and achieve the "three-year plan" and "two rates" goals.

Currently, pregnant women's blood hepatitis B virus load ≥ 2 × 10^5 IU/mL before delivery is the main risk factor that affects transmission prevention and whether infant infection occurs. For pregnant women with high HBV viral load, antiviral therapy during pregnancy can further reduce mother-to-child transmission of HBV. Previous studies have confirmed that tenofovir disoproxil fumarate (TDF) 300mg as a single therapy or combination therapy has good safety and antiviral activity, and can be used as a high viral load for chronic HBV infection as a first-line antiviral treatment for pregnant women. Tenofovir alafenamide (TAF) is a first-line treatment for chronic hepatitis B. Its specification is 25mg. It is an RNA-dependent DNA polymerase inhibitor. The agent is an oral prodrug of tenofovir (TFV), similar to TDF. Because the dosage is much lower than TDF, the incidence of adverse reactions is significantly lower than TDF, but the clinical efficacy is equivalent to TDF. Studies have reported that TAF treatment of HBeAg-positive chronic hepatitis B patients, at 96 weeks HBsAg and HBeAg negative rate, serological conversion rate, ALT normalization rate, etc. were not statistically different from the TDF treatment group. The incidence of ≥ 5% reduction in hip bone and spine bone density, as well as ≥ 5% decrease in estimated glomerular filtration rate (eGFR) from baseline were significantly lower than those in the TDF treatment group. TAF is recommended as the drug of choice for the treatment of chronic hepatitis B.

Extensive past data on pregnant women (over 3,000 exposure outcomes) have shown that there are no malformations or fetal / newborn toxicity associated with TDF. However, no such data exists for TAF. Presently, TAF has been approved by the State Food and Drug Administration (SFDA) and marketed in China in December 2018. SFDA Label has suggested that TAF may be considered during pregnancy if necessary. It has not been reported whether the application of TAF in pregnant women can achieve better effects and safety of mother-to-child transmission prevention, and is the focus of this current study.

This is a multicenter, prospective, triple arm cohort study from the gestational age of 28 weeks in pregnancy to post-partum week 28. The enrollment from 4 centers (Beijing You'an Hospital, Capital Medical University, the Fourth Affiliated Hospital of Harbin Medical University, the third hospital of Qinhuangdao city, Inner Mongolia Tongliao infectious disease hospital) will be caped for sample balance. Consecutive 120 HBeAg-positive and HBV DNA levels ≥ 2 × 10^6 IU/mL pregnant women will be enrolled to receive TAF (25mg oral daily) treatment from the aforementioned 4 centers, consecutive 120 HBeAg-positive and HBV DNA levels ≥ 2 × 10^6 IU/mL pregnant women will be enrolled to receive TDF (300mg oral daily) treatment, and a historical cohort of consecutive highly viremic mothers with HBV DNA levels ≥ 2 × 10^6 IU/mL will be retrospective enrolled as the control group. Patients in the TAF-treated group will receive TAF starting at week 28 of gestation until delivery (if the liver function is abnormal at delivery, ie ALT≥5×ULN, the treatment can be continued according to the wishes of the pregnant woman and the laboratory tests). All infants will receive passive-active immunoprophylaxis. According to the mother's wishes, the mother's milk is collected every day for 5-7 days for TAF concentration determination. In this trial, when the creatinine clearance is less than 15 mL/min, the subjects will discontinue the drug permanently. Subjects with permanent discontinuation (either before or after discontinuation according to the protocol) were followed up every 4 weeks until 16 weeks after discontinuation, or until they received new antiviral treatment. The primary endpoint was the rate of mother-to-child transmission in TAF-treated group compared with control group. The tolerance and safety in TAF-treated group, including congenital malformation rate of infants. The secondary efficacy endpoint was the decrease of HBV DNA level at delivery, the clearance and seroconversion rate of HBsAg or / and HBeAg, ALT normalization and other adverse events of mothers and infants.

For comparison, there will be two comparative arms of mothers whose pregnancies were followed at a single center, Capital Medical University, Beijing Youan Hospital. Arm B will consist of 120 consecutive HBeAg-positive and HBV DNA levels ≥ 2 × 10^6 IU/mL pregnant women enrolled to receive TDF (300mg oral daily) treatment, with all treatment variables constant with the TAF treatment group to act as a control. The TDF treatment for arm B will start at week 28 of gestation until delivery. Arm C will consist of 360 HBeAg-positive and HBV DNA levels ≥ 2 × 10^6 IU/mL pregnant women that did not receive any antiviral treatment during pregnancy. This third group is a historical cohort that will be retrospectively enrolled as an additional comparative arm for further comparison and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Positive Serum tests for both HBsAg and HBeAg
* HBV DNA viremic load ≥ 2 × 10^6 IU/mL
* Mother must be between 20 and 35 years old
* Mother must undergo perinatal testing and delivery at their respective study institution
* Mother must maintain good compliance to study protocols/instructions, as well as any necessary interventions as determined by the local study investigative team.
* Patient must understand and willingly sign an informed consent form provided at enrollment.

Exclusion Criteria:

* Co-infection with the following diseases: HIV-1, Hepatitis A Virus, Hepatitis C Virus, Hepatitis D Virus, Hepatitis E Virus infections or sexually transmitted diseases.
* History of miscarriage or congenital malformations in any previous pregnancy.
* Previous antiviral treatment (except the use of antiviral drugs to prevent MTCT in previous pregnancy and antiviral drugs that have been discontinued for more than 6 months before this pregnancy)
* Previous renal dysfunction
* Liver cancer or liver decompensation
* Creatinine clearance <100 mL / min
* Hypophosphatemia
* Hemoglobin <80g / L
* Neutrophil count <1 × 10 ^ 9 / L
* ALT (U/L) greater than 5x the upper limit of normal
* Total bilirubin > 34.2 umol / L
* Albumin <25g / L
* Any clinical risk/signs of abortion
* Concurrent use of nephrotoxic drugs, steroids, cytotoxic drugs, non-steroidal anti-inflammatory drugs or immune modulators
* Spouse has chronic hepatitis B

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients must be of the female sex, and be pregnant with a child at the time of enrollment.
Study Population: A total of 600 (120 TAF arm A, 120 TDF arm B, 360 arm C) CHB pregnant mothers with high HBV DNA viremic load, i.e. ≥ 2 × 10^6 IU/mL, were included in this study spanning four centers. 120 mothers were prospectively enrolled to take TAF 25 mg per oral at four centers and 120 mothers were prospectively enrolled to take TDF 300mg per oral only at Beijing Youan Hospital, both arms from gestational week 28 until delivery of their infant (if the liver function is abnormal at delivery, ie ALT≥5×ULN, the treatment can be continued according to the wishes of the pregnant woman and the laboratory tests). A historical cohort of 360 consecutive highly viremic mothers who received no antiviral treatment at Beijing Youan Hospital will be retrospective enrolled as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment on the proportion of infants who are infected with hepatitis B at the age of 28 weeks in the two groups | From the date of birth to the age of 24-28 weeks
  Compare MTCT rates between the three study arms and demonstrate non-inferiority in efficacy. MTCT rate is defined as the proportion of infants with serum HBV DNA >20 IU/mL and/or HBsAg positivity at 28 weeks of age.
Assessment on congenital defects and/or malformation rates in each infant group for comparison | From the date of birth to age of 28 weeks
  Congenital defects and/or malformation rates are defined as the proportion of infants with the aforementioned abnormalities discovered during the study period. The proportion of infants who experience congenital defects and/or malformation as determined in all respective groups will be compared.
Tolerability of TDF/TAF therapy: Percentage of mothers who discontinue on TDF/TAF therapy due to the adverse event(s) during the study | Gestational week 28 through delivery of their infant, on average at gestational week 36.
  To evaluate the frequency of treatment discontinuation in patients who could not tolerate TDF/TAF therapy due to adverse event(s) during the study. The proportion of mothers who discontinue TAF therapy as determined in all respective groups will be compared.

SECONDARY OUTCOMES:
Assessment on the reduction of maternal HBV DNA levels at delivery | At delivery
  Assess the percentage of mothers experiencing reduction of maternal HBV DNA levels (IU/mL) > 20,000 IU/mL at delivery when compared to the baseline before initiating TAF/TDF. The proportion of mothers who experience a reduction of maternal HBV DNA levels (IU/mL) > 20,000 IU/mL at delivery as determined in all respective groups will be compared.
Maternal serological outcomes during the study: Percentage of mothers who loss/seroconversion of HBsAg or/and HBeAg during the study | Gestational week 24-28 week to postpartum week 28
  Assess the percentage of mothers who loss/seroconversion of HBsAg or/and HBeAg during the study. Loss is defined by a test showing a negative HBsAg/HBeAg result at the end of the trial, given a positive respective test result at baseline. A seroconversion is defined as a test showing a negative HBsAg and a positive HBsAb result, or a negative HBeAg and a positive HBeAb result at the end of the trial, given a positive HBsAg/HBeAg test result at baseline. The proportion of mothers who experience loss/seroconversion as determined in all respective groups will be compared.
Incidence of Treatment-Emergent Adverse Events in Mothers as Stratified by the CTCAE v 5.0 | Gestational week 24-28 until Postpartum Week 28
  ssess the percentage of Mothers who have adverse events during the study, graded by the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. The proportion of mothers who experience adverse events as determined in all respective groups will be compared.
Incidence of Treatment-Emergent Adverse Events in Infants as Stratified by the CTCAE v 5.0 | At birth until Infant age Week 28
  Assess the percentage of infants who have adverse events during the study, graded by the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. The proportion of infants who experience adverse events as determined in all respective groups will be compared.
Percentage of Mothers with Alanine transferase (ALT) levels within the normal limit | Gestational week 24-28 until Postpartum week 28
  To calculate the percentage of mothers at postpartum 28 weeks whose ALT (U/L) levels stay within the normal limit in response to therapy. The proportion of mothers whose ALT levels who stay within the normal limit as determined in all respective groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongping Duan, MD, Principal Investigator — Capital Medical University, Beijing You'an Hospital; Calvin Q Pan, MD, Study Chair — NYU Langone Health
Locations (4):
- China (4):
  - Beijing You'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Third Hospital of Qinhuangdao City, Qinhuangdao, Hebei
  - Department of Infectious Disease,The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Tongliao Infectious Disease Hospital, Tongliao, Inner Mongolia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jourdain G, Ngo-Giang-Huong N, Harrison L, Decker L, Khamduang W, Tierney C, Salvadori N, Cressey TR, Sirirungsi W, Achalapong J, Yuthavisuthi P, Kanjanavikai P, Na Ayudhaya OP, Siriwachirachai T, Prommas S, Sabsanong P, Limtrakul A, Varadisai S, Putiyanun C, Suriyachai P, Liampongsabuddhi P, Sangsawang S, Matanasarawut W, Buranabanjasatean S, Puernngooluerm P, Bowonwatanuwong C, Puthanakit T, Klinbuayaem V, Thongsawat S, Thanprasertsuk S, Siberry GK, Watts DH, Chakhtoura N, Murphy TV, Nelson NP, Chung RT, Pol S, Chotivanich N. Tenofovir versus Placebo to Prevent Perinatal Transmission of Hepatitis B. N Engl J Med. 2018 Mar 8;378(10):911-923. doi: 10.1056/NEJMoa1708131. PMID 29514030
- [Background] Pan CQ, Duan Z, Dai E, Zhang S, Han G, Wang Y, Zhang H, Zou H, Zhu B, Zhao W, Jiang H; China Study Group for the Mother-to-Child Transmission of Hepatitis B. Tenofovir to Prevent Hepatitis B Transmission in Mothers with High Viral Load. N Engl J Med. 2016 Jun 16;374(24):2324-34. doi: 10.1056/NEJMoa1508660. PMID 27305192
- [Background] Chen HL, Lee CN, Chang CH, Ni YH, Shyu MK, Chen SM, Hu JJ, Lin HH, Zhao LL, Mu SC, Lai MW, Lee CL, Lin HM, Tsai MS, Hsu JJ, Chen DS, Chan KA, Chang MH; Taiwan Study Group for the Prevention of Mother-to-Infant Transmission of HBV (PreMIT Study); Taiwan Study Group for the Prevention of Mother-to-Infant Transmission of HBV PreMIT Study. Efficacy of maternal tenofovir disoproxil fumarate in interrupting mother-to-infant transmission of hepatitis B virus. Hepatology. 2015 Aug;62(2):375-86. doi: 10.1002/hep.27837. Epub 2015 May 13. PMID 25851052
- [Background] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- [Background] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- [Derived] Zou H, Zhu L, Cao L, Suo S, Zhu Y, Wang Y, Dong J, Han B, Duan Z, Chen Y, Pan CQ. Vertical Transmission in Mothers Taking TAF With Exceptionally High Viral Load. J Viral Hepat. 2025 Mar;32(3):e70000. doi: 10.1111/jvh.70000. PMID 39953819